CLINICAL TRIAL: NCT00781443
Title: A Phase II, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MILR1444A in the Prevention of Allergen-Induced Airway Obstruction in Adults With Mild Allergic Asthma
Brief Title: A Study to Evaluate MILR1444A in the Prevention of Allergen-Induced Airway Obstruction in Adults With Mild Allergic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILR4544g
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Last update posted 2010-05-06 (Estimated); Status verified 2010-05

CONDITIONS: Allergic Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- A (Experimental)
  Interventions: Drug: lebrikizumab (MILR1444A)
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lebrikizumab (MILR1444A) — Repeating subcutaneous injection
  Arms: A
Drug: placebo — Repeating subcutaneous injection
  Arms: B

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study designed to demonstrate the safety and efficacy of MILR1444A compared with placebo in reducing the airway reaction to an inhaled aeroallergen solution in adult patients with mild allergic asthma. The study will randomize approximately 24 patients at five study centers. In the event of patient discontinuation from the study, additional patients may be enrolled at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for the diagnosis of allergic asthma
* Diagnosis of asthma ≥ 6 months
* Currently treated with only intermittent short-acting inhaled β-adrenergic agonists
* Body weight between 40-120 kg
* Normal chest X-ray within 2 years of screening

Exclusion Criteria:

* Require daily controller medication for asthma
* History of hypersensitivity to the study drug or to drugs with similar chemical structures or to any ingredients, including excipients of the study medication or drugs related to MILR1444A (e.g., monoclonal antibodies, polyclonal gamma globulin)
* Documented medical history of anaphylaxis
* Immunotherapy currently or within the past 3 months prior to screening
* Lung disease other than mild allergic asthma
* Previous treatment with other investigational drugs within 30 days or 5 half-lives prior to the screening visit, whichever is longer
* Pregnant or lactating
* Significant concurrent medical illness other than asthma
* Clinically significant abnormality on ECG at the screening visit
* Smoked in the previous 6 months or have a history of smoking more than 10 pack-years
* History of helminthic infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Late asthmatic response (LAR) | Day 92

SECONDARY OUTCOMES:
Early asthmatic response (EAR) | Day 92

CONTACTS AND LOCATIONS:
Overall Officials: Edward Conner, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Scheerens H, Arron JR, Zheng Y, Putnam WS, Erickson RW, Choy DF, Harris JM, Lee J, Jarjour NN, Matthews JG. The effects of lebrikizumab in patients with mild asthma following whole lung allergen challenge. Clin Exp Allergy. 2014 Jan;44(1):38-46. doi: 10.1111/cea.12220. PMID 24131304